CLINICAL TRIAL: NCT02529644
Title: Assessing HIV Screening in African American Churches
Brief Title: Church-based HIV Screening: Taking It to the Pews
Acronym: TIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: City of Kansas City Missouri Health Department (Unknown); Kansas City CARE Clinic (Unknown); RAND (Other); Children's Mercy Hospital Kansas City (Other); Caanon Worship Center (Unknown); Christian Fellowship Baptist Church (Unknown); Friendship Baptist Church (Unknown); JayDoc Free Clinic (Unknown); Metropolitan Spiritual Church of Christ (Unknown); NBC Community Development Corporation (Unknown); Concord Fortress of Hope Church (Unknown); Victorious Life Church (Unknown); Calvary Community Outreach Network (Unknown)
Responsible Party: Principal Investigator, Jannette Berkley-Patton, Associate Professor of Biomedical and Health Informatics, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 13-926
Record Dates: First submitted 2015-08-06; First posted 2015-08-20 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: HIV
Keywords: HIV Screening; African American; Church
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comparison (Standard Information Arm) (Active Comparator): The comparison/standard information churches will receive standard multilevel HIV education information that is similar in type to those provided to the intervention churches. These churches will receive: a) non-tailored project materials (videos, brochures) collected from health organizations and b) standard, non-tailored activities (e.g., community-based HIV testing events) coordinated by their church liaisons. These churches will receive all Taking It to the Pews HIV Tool Kit materials after the completion of 12-month assessments.
  Interventions: Behavioral: Taking It to the Pews (Comparison)
- Intervention (Experimental): Taking It to the Pews (TIPS) will be delivered through church-based multilevel (community, church-wide, ministry group, interpersonal/individual) activities by trained church leaders using religiously/ culturally-tailored study materials packaged in a TIPS HIV Tool Kit and following a scripted, study implementation manual.
  Interventions: Behavioral: Taking It to the Pews (Experimental)

INTERVENTIONS:
Behavioral: Taking It to the Pews (Comparison) — Pastors and Health Action Team members will be trained and receive manualized pastor/church liaison trainings on study procedures, HIV basics and local resources and coordination of HIV screening events. Comparison churches will receive: a) non-tailored project materials (videos, brochures) collected from health organizations and b) standard, non-tailored activities (e.g., community-based HIV testing events) coordinated by their church liaisons. The comparison churches will offer 3 HIV screening events and deliver 1-2 standard materials per month for the 12 month study period. All comparison churches will receive all Taking It to the Pews HIV Tool Kit materials after the completion of 12-month assessments.
  Other Names: TIPS
  Arms: Comparison (Standard Information Arm)
Behavioral: Taking It to the Pews (Experimental) — Pastors and Health Action Team members will be trained in treatment implementation procedures using the scripted, study implementation manual. Intervention churches will receive the TIPS HIV Tool Kit, including a study manual. These churches will hold a Kick-off event, where tools will be distributed, and motivational strategies implemented. After the Kick-off, liaisons will deliver 1-2 Tool Kit materials/activities per month through targeted multilevel church activities minimum of 24 tools over the 12 month study period. Two additional HIV screening events will be planned (one for community members) and will be open to all persons seeking screening, including study nonparticipants. Both groups will receive manualized pastor/church liaison trainings on study procedures, HIV basics and local resources and coordination of HIV screening events.
  Other Names: TIPS
  Arms: Intervention

SUMMARY:
The primary aim of this study is to fully test a culturally/religiously-tailored, church-based HIV screening intervention (TIPS) against a standard HIV information intervention on HIV screening rates at 6 and 12 months with adult African American church members and community members who use church outreach services. Our secondary outcome is to reduce sexual risk behaviors with this same population.

DETAILED DESCRIPTION:
The primary aim of this study is to fully test a culturally/religiously-tailored, church-based HIV screening intervention against a standard HIV information intervention on HIV screening rates at 6 and 12 months with adult AA church members and community members who use church outreach services. In this two-arm clustered, randomized community trial, churches will be matched on SES, membership size, and denomination, then randomized to treatment condition. It is projected that 14 churches (7 churches per arm; 110 church and community members per church; 1,540 participants total) will be required to detect significant increases in HIV screening in the intervention arm. Intervention content is guided by the Theory of Planned Behavior (TPB). Intervention delivery will be guided by a Community Engagement and Social-Ecological approach. This approach includes church leaders delivering culturally/religiously-appropriate HIV education and screening materials (e.g., sermon guides, HIV screening testimonials, church bulletins) and activities (e.g., pastors modeling receipt of HIV screening, HIV screening events) from a church-based HIV Tool Kit through multilevel church outlets (community-wide, church-wide services, ministry and outreach groups, individual) to increase intervention reach and dosage. It was hypothesized that this church-based HIV screening intervention will significantly increase HIV screening rates vs a standard HIV information intervention in AA church-populations at 6 and 12 months. The role of potential mediators and moderators related to receipt of HIV screening will be evaluated and a process evaluation to determine modifiable implementation fidelity, facilitators, barriers, and costs related to increasing church-based HIV testing rates will be conducted. This intervention study could provide an effective, scalable model for HIV screening interventions in AA churches.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be: aged 18 to 64; willing to participate in 3 surveys after church services or church outreach activities
* Willing to provide contact information (two phone numbers, mailing and email address, phone numbers for two persons with whom they have ongoing contact)
* Attend church at least once a month or use church outreach services, such as food and clothing programs, at least 4 times per year.

Exclusion Criteria:

* Minors 18 and under are intentionally excluded since the intervention study has been designed specifically for adults with information of how HIV affects the African American adult population.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1540 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported Receipt of HIV Screening | Baseline
  This measure is self-reported receipt of HIV screening received in last 12 months
Self-reported Receipt of HIV Screening | 6 months
  This measure is self-reported receipt of HIV screening recieved in last 12 months
Self-reported Receipt of HIV screening | 12 months
  This measure is self-reported receipt of HIV screening received in last 12 months

SECONDARY OUTCOMES:
HIV Sexual Risk Behavior Score | Baseline
  HIV sexual risk behavior will be assessed as a composite measure: a) if participant had vaginal, oral, or anal sex with (No=0, Yes=1); b) the number of men and the number of women they had sex with, recoded as 1 to 5 sex partners=1 and 6 or more sex partners=2; and c) how often they or partner(s)/spouse used condoms or barriers (Always=0, Usually=1, Sometimes=2, or Never=3) within last 12 months. Higher scores indicate more sexual risk (range 0-8).
HIV Sexual Risk Behavior Score | 6 months
  HIV sexual risk behavior will be assessed as a composite measure: a) if participant had vaginal, oral, or anal sex with (No=0, Yes=1); b) the number of men and the number of women they had sex with, recoded as 1 to 5 sex partners=1 and 6 or more sex partners=2; and c) how often they or partner(s)/spouse used condoms or barriers (Always=0, Usually=1, Sometimes=2, or Never=3) within last 12 months. Higher scores indicate more sexual risk (range 0-8).
HIV Sexual Risk Behavior Score | 12 months
  HIV sexual risk behavior will be assessed as a composite measure: a) if participant had vaginal, oral, or anal sex with (No=0, Yes=1); b) the number of men and the number of women they had sex with, recoded as 1 to 5 sex partners=1 and 6 or more sex partners=2; and c) how often they or partner(s)/spouse used condoms or barriers (Always=0, Usually=1, Sometimes=2, or Never=3) within last 12 months. Higher scores indicate more sexual risk (range 0-8).

CONTACTS AND LOCATIONS:
Overall Officials: Jannette Y. Berkley-Patton, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- University of Missouri-Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Berkley-Patton J, Thompson CB, Bauer AG, Berman M, Christensen K, Bradley-Ewing A, Goggin K, Catley D, Williams E, Wainright C, Derose KP, Geyer A, Thompson F, Dennis L, Smith S, Allsworth JE. HIV Testing in African American Churches: Results from the Taking It to the Pews Cluster-Randomized Trial. AIDS Behav. 2026 Jan;30(1):118-129. doi: 10.1007/s10461-025-04852-2. Epub 2025 Aug 29. PMID 40880008

DOCUMENTS (3):
  • Informed Consent Form (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02529644/ICF_000.pdf
  • Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT02529644/SAP_001.pdf
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT02529644/Prot_002.pdf